CLINICAL TRIAL: NCT03337919
Title: A Phase II Study of Nivolumab Monotherapy in Patients With Relapsed/Refractory Hodgkin Lymphoma Fit for Autologous Stem Cell Transplant Who Fail to Reach Complete Metabolic Remission After First or Second Line Salvage Therapy
Brief Title: ANIMATE: Phase II Study of Nivolumab Monotherapy for Relapsed/Refractory Hodgkin Lymphoma
Acronym: ANIMATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/15/0515; CA-209-445 (Other Grant/Funding Number: Bristol-Myers Squibb); 2017-002544-32 (EudraCT Number)
Record Dates: First submitted 2017-10-26; First posted 2017-11-09 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hodgkin Lymphoma
Keywords: Nivolumab
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a single-arm, phase II, multi-centre study. It will use an Ahern single stage design with independent trials steering committee review to monitor for safety and efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab (Experimental): Up to 8 x 2-weekly cycles of nivolumab 240mg IV. Interim PET-CT scan to be performed after 4 cycles, and centrally reviewed. Patients will stop treatment after 4 cycles if they have complete metabolic response or progressive metabolic disease. If they have partial metabolic response or stable disease, they will continue to 8 cycles.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Up to 8 cycles of nivolumab
  Other Names: Opdivo®

SUMMARY:
This is a single-arm, phase II, multi-centre study of the safety and efficacy of the PD-1 inhibitor, nivolumab, as second-line or third-line salvage therapy as a bridge to stem cell transplant (SCT) in relapsed/ refractory classical Hodgkin lymphoma patients not achieving a complete metabolic response (CMR) on FDG-PET-CT scan after first or second line salvage therapy.

DETAILED DESCRIPTION:
This is a single-arm, phase II, multi-centre study of the safety and efficacy of the programmed cell death protein 1 (PD-1) inhibitor, nivolumab, as second-line or third-line salvage therapy, and in particular as a bridge to stem cell transplant (SCT) in relapsed/ refractory classical Hodgkin lymphoma patients not achieving a complete metabolic response (CMR) on fluorodeoxyglucose positron emission tomography (FDG-PET) scan post first or second line salvage therapy.

Approximately 120 patients with relapsed/refractory classical Hodgkin lymphoma will be registered while undergoing first or second line salvage therapy (first line is preferred).

Patients will have a centrally reviewed PET CT scan after first or second line salvage therapy. Those with complete metabolic response (CMR) on PET CT scan (Deauville score 1-3) will not be eligible for trial treatment. They will be followed up for trial data collection purposes, and further management will be at their treating clinician's discretion.

Patients achieving less than CMR on central review of FDG-PET (Deauville score 4-5) will be eligible to receive up to 8 x 2-weekly nivolumab infusions. 30 patients will be treated on the trial.

After 4 courses of nivolumab, patients will have an additional centrally reviewed PET-CT scan (PET4). Patients achieving CMR will stop trial treatment, and enter follow up. Further treatment will be at their clinician's discretion but is likely to be stem cell transplant (SCT). Patients with partial metabolic response (PMR) or stable disease (SD) on PET4 will receive a further 4 cycles of nivolumab, again followed by a centrally reviewed PET-CT scan (PET8) to assess final response.

Further management after PET8 will be at the discretion of the treating clinician, although it is anticipated that those with CMR or PMR will proceed to SCT. If PET8 shows less than CMR (i.e. PMR or SD), patients who consent will have a further biopsy to exclude false positive PET signal; this will be centrally reviewed.

Patients with progressive metabolic disease (PMD) on nivolumab at any point will stop trial treatment. If a repeat biopsy is obtained to confirm progressive disease histologically, the biopsy material will be centrally reviewed.

Patients will be followed up for a minimum of 3 years.

ELIGIBILITY:
Inclusion criteria for study registration:

1. Age 16 or over
2. Primary refractory classical Hodgkin lymphoma or classical Hodgkin lymphoma in first relapse
3. About to receive or receiving first or second line salvage therapy (up to a maximum of 14 days after last treatment)
4. Fit for autologous stem cell transplantation
5. Written informed consent
6. Willing to comply with the contraceptive requirements of the trial

Exclusion criteria for study registration:

1. Nodular lymphocyte predominant Hodgkin lymphoma
2. Women who are pregnant or breastfeeding
3. History of colitis, inflammatory bowel disease or pneumonitis
4. Patients with autoimmune disorders, except patients with vitiligo, diabetes mellitus type 1, hypo- and hyperthyroidism not requiring immunosuppressive therapy
5. Known history of hepatitis B or C infection
6. Known HIV infection
7. History of allergy (including severe/life threatening skin reaction) to monoclonal antibodies, anaphylaxis or uncontrolled allergy
8. Major surgery within 4 weeks prior to registration
9. Myocardial infarction, unstable angina, coronary artery bypass graft, cerebrovascular accident or transient ischaemic attack within the past 6 months
10. Non-haematological malignancy within the past 3 years (with some exceptions - listed in protocol)

Inclusion criteria for trial treatment:

1. Has received 2 cycles of first or second line salvage chemotherapy
2. PET positive (Deauville score 4 or 5) after first or second line salvage chemotherapy
3. Fit for further salvage chemotherapy
4. ECOG performance status 0-1
5. Creatinine clearance >30ml/min calculated by Cockcroft-Gault formula
6. Bilirubin <1.5 x ULN, ALT/AST <2.5 x ULN
7. Adequate bone marrow function (Hb >80g/l, Platelets >50 x 10^9/l, neutrophils >1.0 x 10^9/l)

Exclusion criteria for trial treatment:

1. Deauville score 1-3 after first or second line salvage chemotherapy
2. Positive serology for hepatitis B or C (some exclusions apply - see protocol)
3. Active infection requiring systemic therapy
4. Ongoing requirement for immunosuppressive therapy, apart from inhaled, intranasal, topical corticosteroids or systemic corticosteroids at low doses (≤10mg prednisolone per day, or the equivalent)
5. Corticosteroids at a dose of more than 10mg per day prednisolone or equivalent within 7 days prior to response PET-CT. NOTE: corticosteroids can be used AFTER a positive PET-CT scan for symptomatic disease but must be weaned to a dose of prednisolone ≤10mg/day or less (or equivalent) at least 7 days prior to starting nivolumab.
6. Treatment with any investigational agent within 28 days prior to planned start of nivolumab
7. Ongoing grade 2-4 non-haematological toxicities related to prior Hodgkin lymphoma treatments, with the exception of alopecia and grade 2 fatigue
8. Pregnant or breastfeeding women

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) by PET-CT scan following 4-8 cycles of nivolumab | 4 months
  Rate of patients achieving complete metabolic response (CMR) on PET-CT scan following 4 or 8 cycles of nivolumab

SECONDARY OUTCOMES:
Progression-free survival | 1 year
  Progression-free survival at 1 year; also to be analysed stratified by partial metabolic response vs complete metabolic response.
Overall survival | 1 year
  Overall survival at 1 year; also to be analysed stratified by partial metabolic response (PMR) vs complete metabolic response (CMR).
Proportion of patients progressing to stem cell transplant | 1 year
  Proportion of patients progressing to autologous or allogeneic stem cell transplant
Adverse events [Safety and toxicity of nivolumab] | 3 years
  Adverse events and serious adverse events occurring in patients treated with nivolumab, in particular autoimmune toxicity
Transplant-related mortality | 3 years
  Proportion of patients treated with nivolumab that subsequently die of transplant-related causes
Transplant-related morbidity | 3 years
  Proportion of patients treated with nivolumab that go on to suffer serious complications of allogeneic transplant (grade 3-4 graft-versus-host disease, hyperacute graft-versus-host disease and steroid-responsive febrile syndrome)

OTHER OUTCOMES:
Biopsy-negative PMR rate | 4 months
  Correlation of PET positive disease with histological evidence of disease on post-treatment repeat biopsy to establish biopsy negative PMR rate (subject to patient consent)
Serological biomarkers of response to nivolumab | 5 months
  Correlation of disease response with serological markers such as serum Thymus and activation-regulated chemokine (TARC) levels
Immunological biomarkers of response to treatment | 4 months
  Evaluate the correlation between response to nivolumab and biological parameters e.g. PD-L1 expression on Reed Sternberg cells

CONTACTS AND LOCATIONS:
Overall Officials: Graham Collins, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (10):
- United Kingdom (10):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Norfolk & Norwich University Hospital, Norwich, Norfolk
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Leicester Royal Infirmary, Leicester
  - St Bartholomew's Hospital, London
  - Guy's Hospital, London
  - St George's Hospital, London
  - The Royal Marsden Hospital, London
  - The Christie Hospital, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CR UK & UCL Cancer Trials Centre — http://www.ctc.ucl.ac.uk/